CLINICAL TRIAL: NCT00212693
Title: Controlled Study of ONO-2506PO in Patients With Parkinson's Disease in Japan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-2506PO-03
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Parkinson's Disease
Keywords: ONO-2506PO, Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

INTERVENTIONS:
Drug: ONO-2506PO

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ONO-2506PO in patients with Parkinson's Disease

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Parkinson's disease
2. Stage 2 - Stage 4 of revised Hoehn & Yahr severity score
3. Taking L-dopa/DCI without changing dose and regimen
4. Having motor complication
5. Other inclusion criteria as specified in the study protocol

Exclusion Criteria:

1. Previous participation in ONO-2506PO or ONO-2506 protocol
2. Previous brain surgery for Parkinson's disease
3. Presence or history of serious cardiac disease
4. Other exclusion criteria as specified in the study protocol

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165
Dates: Start 2004-01; Primary Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's disease rating scale (Part III)

SECONDARY OUTCOMES:
Unified Parkinson's disease rating scale (Part I, II, IV and total), revised Hoehn & Yahr severity score and off time

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Development Planning, Study Director — Ono Pharmaceutical Co. Ltd